CLINICAL TRIAL: NCT02772874
Title: Clinical, Anatomic, and Physiologic Characteristics of Fecal Incontinence Subtypes in Women With Pelvic Floor Disorders
Brief Title: Fecal Incontinence Subtypes in Women With Pelvic Floor Disorders
Acronym: FIST
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 820286
Record Dates: First submitted 2015-02-03; First posted 2016-05-16 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; severity; ultrasound; anorectal manometry; classification
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urge-predominant: All subjects who report fecal incontinence that is primarily urge-predominant will undergo self-administered questionnaires, pelvic examination, endoanal ultrasound, and anorectal manometry.
  Interventions: Other: No intervention
- Passive-predominant: All subjects who report fecal incontinence that is primarily passive-predominant will undergo self-administered questionnaires, pelvic examination, endoanal ultrasound, and anorectal manometry.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Fecal incontinence (FI) is clinically subtyped as urge FI and passive FI based on symptoms, however the pathophysiologic significance of this subtyping is not known. FI is commonly encountered in women with pelvic floor disorders. This study aims to compare characteristics of clinical severity, quality of life, anatomy, and physiology of urge FI versus passive FI. Urogynecology patients greater than age 18 with FI at least monthly over the last 3 months will be recruited for participation. Participants will be divided into urge FI subtype and passive FI subtype. Participants will complete validated questionnaires on clinical severity and quality of life, both as related to FI and general heath. Participants will undergo pelvic examination, endoanal ultrasound and anorectal manometry for evaluation of anatomic and physiologic pathology. Results between both groups will be compared. The investigators hypothesize that clinical, anatomic, and physiologic characteristics differ between urge-predominant fecal incontinence and passive-predominant fecal incontinence in women with pelvic floor disorders.

DETAILED DESCRIPTION:
Fecal incontinence greatly affects quality of life and can negatively impact an individual's activity level, body image, and likelihood of institutionalization. Female sex and advancing age are known independent risk factors for fecal incontinence. Among community dwelling adults, the prevalence of fecal incontinence has ranged from 0.4 to 18 percent. Prevalence rates of fecal incontinence are even higher in women with pelvic floor disorders, reaching up to 41%, illustrating the large bearing on quality of life of this patient population.

Fecal incontinence can be subtyped into three clinical subtypes: urge fecal incontinence, passive fecal incontinence, and fecal seepage. Urge incontinence refers to loss of fecal matter in spite of active attempts to retain contents; passive incontinence refers to involuntary loss of stool without awareness. Despite the clinical distinction of fecal incontinence subtypes, the pathophysiology of these subtypes is not known. Existing practice guidelines recommend categorizing patients into these subtypes, evaluating symptom severity by patient-reported outcomes, and assessing function of the anorectal complex with imaging and physiologic tests to best tailor management options. Although the framework for subtyping fecal incontinence exists, specific associations between subtypes and clinical, anatomic, and physiologic findings in women with pelvic floor disorders are not well delineated. Further characterizing the subtypes in relation to specific clinical, anatomic, and physiologic findings may allow us to better approach the treatment of women with fecal incontinence.

Our comparison of the two fecal incontinence subtypes, urge-predominant fecal incontinence and passive fecal incontinence, will be evaluated for clinical severity, impact on quality of life, and anatomic and physiologic characteristics using validated instruments.

Primary Aim:

To compare the severity of urge fecal incontinence versus passive fecal incontinence in women with pelvic floor disorders.

Secondary Aims:

1. To compare anatomic characteristics in urge fecal incontinence versus passive fecal incontinence in women with pelvic floor disorders.
2. To compare physiologic characteristics in urge fecal incontinence versus passive fecal incontinence in women with pelvic floor disorders.
3. To compare quality of life characteristics in urge fecal incontinence versus passive fecal incontinence in women with pelvic floor disorders.
4. To compare anorectal manometry results and patient preference of testing performed in the left lateral position versus dorsal lithotomy position.

Null Hypothesis: Clinical, anatomic, and physiologic characteristics do not differ between urge-predominant fecal incontinence and passive-predominant fecal incontinence in women with pelvic floor disorders.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than age 18 with fecal incontinence at least monthly over the last 3 months

Exclusion Criteria:

* Malignancy
* Fistula
* Rectal prolapse
* Prior colorectal surgery
* Prior radiation
* Fecal impaction
* Sole flatal incontinence
* Neurologic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women greater than age 18 with fecal incontinence at least monthly over the last 3 months being evaluated in the Urogynecology office setting.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Fecal incontinence severity as measured by mean Vaizey score | Participants will be assessed for this outcome at their sole primary visit and data will be presented approximately 1 year later.
  Vaizey score range 0 to 24

SECONDARY OUTCOMES:
Anal anatomy patency as measured by mean anal sphincter complex thickness (millimeters). | Participants will be assessed for this outcome at their sole primary visit and data will be presented approximately 1 year later.
  Internal anal sphincter thickness (millimeters) and external anal sphincter thickness (millimeters) at 12, 3, 6, 9 o'clock.
Anal anatomy patency as measured by presence or absence of defects using endoanal ultrasound. | Participants will be assessed for this outcome at their sole primary visit and data will be presented approximately 1 year later.
  The presence of defects anywhere along internal anal sphincter or external anal sphincter will be measured as present or absent.
Anal function as measured by the anorectal manometry measurements (see description below). | Participants will be assessed for this outcome at their sole primary visit and data will be presented approximately 1 year later.
  Mean anal resting pressure at high pressure zone (mmHg), mean anal squeeze pressure (mmHg), mean anal squeeze duration (seconds), mean rectal first sensation capacity (cc), mean rectal normal urge capacity (cc), mean rectal strong urge capacity (cc), and mean maximum tolerated volume capacity (cc).
Rectal function as measured by the anorectal manometry measurements (see description below). | Participants will be assessed for this outcome at their sole primary visit and data will be presented approximately 1 year later.
  Mean rectal first sensation capacity (cc), mean rectal normal urge capacity (cc), mean rectal strong urge capacity (cc), and mean maximum tolerated volume capacity (cc).

CONTACTS AND LOCATIONS:
Overall Officials: Avita K Pahwa, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Division of Urogynecology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bharucha AE, Zinsmeister AR, Locke GR, Seide BM, McKeon K, Schleck CD, Melton LJ. Prevalence and burden of fecal incontinence: a population-based study in women. Gastroenterology. 2005 Jul;129(1):42-9. doi: 10.1053/j.gastro.2005.04.006. PMID 16012933
- [Background] Nelson R, Norton N, Cautley E, Furner S. Community-based prevalence of anal incontinence. JAMA. 1995 Aug 16;274(7):559-61. PMID 7629985
- [Background] Macmillan AK, Merrie AE, Marshall RJ, Parry BR. The prevalence of fecal incontinence in community-dwelling adults: a systematic review of the literature. Dis Colon Rectum. 2004 Aug;47(8):1341-9. doi: 10.1007/s10350-004-0593-0. PMID 15484348
- [Background] Bezerra LR, Vasconcelos Neto JA, Vasconcelos CT, Karbage SA, Lima AC, Frota IP, Rocha AB, Macedo SR, Coelho CF, Costa MK, Souza GC, Regadas SM, Augusto KL. Prevalence of unreported bowel symptoms in women with pelvic floor dysfunction and the impact on their quality of life. Int Urogynecol J. 2014 Jul;25(7):927-33. doi: 10.1007/s00192-013-2317-2. Epub 2014 Feb 22. PMID 24562788
- [Background] Rao SS; American College of Gastroenterology Practice Parameters Committee. Diagnosis and management of fecal incontinence. American College of Gastroenterology Practice Parameters Committee. Am J Gastroenterol. 2004 Aug;99(8):1585-604. doi: 10.1111/j.1572-0241.2004.40105.x. No abstract available. PMID 15307881
- [Background] Rao SS. Pathophysiology of adult fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S14-22. doi: 10.1053/j.gastro.2003.10.013. PMID 14978634
- [Derived] Pahwa AK, Khanijow KD, Harvie HS, Arya LA, Andy UU. Comparison of Patient Impact and Clinical Characteristics Between Urgency and Passive Fecal Incontinence Phenotypes. Female Pelvic Med Reconstr Surg. 2020 Sep;26(9):570-574. doi: 10.1097/SPV.0000000000000603. PMID 29979355